CLINICAL TRIAL: NCT03306732
Title: Thiamine Supplementation in High Risk Cardiac Surgery Patients
Acronym: APPLY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Efremov Sergey, MD PHD Principal Investigator, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2017-09-19; First posted 2017-10-11 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Cardiac Surgery
Keywords: Thiamine; Thiamine Supplementation; Vasoplegia Syndrome; Inotropic support; Cardiac surgery; Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — thiamine hydrochloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thiamine group (Active Comparator)
  Interventions: Drug: Thiamine hydrochloride (200mg) dissolved in 100 ml of normal saline
- Placebo group (Placebo Comparator)
  Interventions: Drug: Normal saline (100ml)

INTERVENTIONS:
Drug: Thiamine hydrochloride (200mg) dissolved in 100 ml of normal saline — * After anesthesia induction
  * After separation from CPB
  * On the evening of the day of surgery (22:00)
  * On POD 1 twice a day at 8:00 and 22:00
  * On POD 2 twice a day at 8:00 and 22:00 (if patient is still in ICU)
  * On POD 3 twice a day at 8:00 and 22:00 (if patient is still in ICU)
  Arms: Thiamine group
Drug: Normal saline (100ml) — * After anesthesia induction
  * After separation from CPB
  * On the evening of the day of surgery (22:00)
  * On POD 1 twice a day at 8:00 and 22:00
  * On POD 2 twice a day at 8:00 and 22:00 (if patient is still in ICU)
  * On POD 3 twice a day at 8:00 and 22:00 (if patient is still in ICU)
  Arms: Placebo group

SUMMARY:
This pilot trial will evaluate the ability of thiamine to affect on postoperative vasoplegia in high risk cardiac surgery patients

DETAILED DESCRIPTION:
Thiamine has a pivotal role and is an essential cofactor for pyruvate dehydrogenase activity. Widely known wet beri-beri is developed due to thiamine deficiency and characterized by vasodilatory shock and despaired oxygen extraction leading to kidney, heart and central nervous system dysfunction. Thiamine deficiency is often underestimated and even in primary absence of vitamin B1 deficiency, high-consumptive state of many critical illness and cardiac surgery itself can lead to its lack. Reported that in patients on chronic dialysis and patients with AKI requiring RRT thiamine deficiency is a usual finding. In cross-sectional observational study it has been shown that up to 33% of patients with a diagnosis of congestive heart failure (CHF) had thiamine deficiency due to chronic loop diuretic use. Also reported that 96% of patients (21 of 23) with heart failure receiving loop diuretic therapy (daily dose: 80-240 mg furosemide) developed thiamine deficiency. In prospective observational trial it has been shown that plasma thiamine levels were decreased after CABG surgery.

In a secondary analysis of a randomized, double-blind, placebo-controlled trial conducted in septic patients, thiamine supplementation showed highly-promising renal protective effect. Need for RRT was 8 patients (21%) in placebo group and 1 patient (3%) in thiamine group (p=0.04).

On the other hand it was unable to show any benefit of thiamine supplementation in patients undergoing CABG surgery. Although, postoperative oxygen consumption was significantly increased among patients receiving thiamine.

Nevertheless, existing evidence suggests that thiamine supplementation might be an attractive strategy in counteracting organ dysfunction and thus morbidity and mortality in high-risk cardiac surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Valve surgery + CABG that required cardiac surgery with CPB
* Aged 18 years or older
* Signed informed consent

Exclusion Criteria:

* Emergency surgery
* Chronic kidney disease of G4-G5 categories according to KDIGO criteria (at least one of the following present for > 3 months: glomerular filtration rate ≤ 29 ml/min/1.73 m2, history of kidney transplantation)
* Known allergy to thiamine
* Pregnancy
* Current enrollment into another RCT (in the last 30 days)
* Previous enrollment and randomisation into the APPLY trial
* Administration of thiamine in the previous 30 day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 8 month
  Recruitment of trial patients: successful recruitment is defined as 2 patients per week on average
Compliance with the protocol | 8 month
  Successful compliance with protocol is defined as ≥ 90% of prescribed intervention being administered across all patients

SECONDARY OUTCOMES:
Vasoinotropic score | 3 days
  dosage of vasoinotropic agents and total vasopressor/norepinephrine equivalent dose
Peak lactate level after CPB weaning to 48 hours | 48 hours
The value of postoperative peak serum creatinine concentration during 3 postoperative days | 3 days
The incidence of acute kidney injury (AKI) according to "Kidney Disease: Improving Global Outcomes (KDIGO) criteria" during ICU stay | 30 days
The daily incidence of cardiovascular and renal dysfunction according to Sequential Organ Failure Assessment (SOFA) score during 48 hours postoperatively | 48 hours
Rates of postoperative complications | 30 days
Incidence of Treatment-Emergent Adverse Events | 30 days
  The safety of high dose IV thiamine supplementation will be evaluated by comparison of adverse, serious adverse events and routinely assessed biochemical parameters (i.e. complete blood count, coagulation parameters, standard biochemistry, etc.)
Availability of data needed | 8 month
  We expect that loss of follow up will not exceed 5% and data loss less than 10%
7-day all-cause mortality (or mortality at any time during the first hospitalization) | 7 days
30-day all-cause mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin Research Institute of Pathology of Circulation, Novosibirsk, Russia

REFERENCES:
- [Background] Wiesen P, Van Overmeire L, Delanaye P, Dubois B, Preiser JC. Nutrition disorders during acute renal failure and renal replacement therapy. JPEN J Parenter Enteral Nutr. 2011 Mar;35(2):217-22. doi: 10.1177/0148607110377205. PMID 21378251
- [Background] Seligmann H, Halkin H, Rauchfleisch S, Kaufmann N, Motro M, Vered Z, Ezra D. Thiamine deficiency in patients with congestive heart failure receiving long-term furosemide therapy: a pilot study. Am J Med. 1991 Aug;91(2):151-5. doi: 10.1016/0002-9343(91)90007-k. PMID 1867241
- [Background] Donnino MW, Cocchi MN, Smithline H, Carney E, Chou PP, Salciccioli J. Coronary artery bypass graft surgery depletes plasma thiamine levels. Nutrition. 2010 Jan;26(1):133-6. doi: 10.1016/j.nut.2009.06.004. PMID 20005469
- [Background] Andersen LW, Holmberg MJ, Doherty M, Khabbaz K, Lerner A, Berg KM, Donnino MW. Postoperative Lactate Levels and Hospital Length of Stay After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2015 Dec;29(6):1454-60. doi: 10.1053/j.jvca.2015.06.007. Epub 2015 Jun 6. PMID 26456273

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT03306732/Prot_SAP_000.pdf